CLINICAL TRIAL: NCT06822270
Title: Evaluation of Different Surgical Modalities in the Management of Pelvi-ureteric Junction Obstruction: a Randomized Controlled Trial
Brief Title: Different Surgical Modalities in the Management of Pelvi-ureteric Junction Obstruction
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Mohamed Gamil Ahmed Saleh, Dr, Al-Azhar University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MD/AZ.AST/AIP029/21/186/3/2018
Record Dates: First submitted 2024-12-28; First posted 2025-02-12 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2025-02

CONDITIONS: Pelvi-ureteric Junction Obstruction
MeSH Terms: conditions — Multicystic renal dysplasia, bilateral | interventions — Conversion to Open Surgery

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Open Pyeloplasty Group (Active Comparator): This group underwent traditional open surgical methods for treating Pelvi-ureteric Junction Obstruction.
  Interventions: Procedure: open surgery
- Laparoscopic Pyeloplasty Group (LP) (Experimental): This group was treated using minimally invasive laparoscopic techniques.
  Interventions: Procedure: Laparoscopic Pyeloplasty

INTERVENTIONS:
Procedure: open surgery — open surgical methods for treating Pelvi-ureteric Junction Obstruction
  Arms: Open Pyeloplasty Group
Procedure: Laparoscopic Pyeloplasty — minimally invasive laparoscopic techniques.
  Arms: Laparoscopic Pyeloplasty Group (LP)

SUMMARY:
The study compared open pyeloplasty (OP) and laparoscopic pyeloplasty (LP) for treating Pelvi-ureteric Junction Obstruction (PUJO) in 40 patients.

ELIGIBILITY:
Inclusion Criteria:

* Age between 7 months and 60 years. Diagnosed with Pelvi-ureteric Junction Obstruction (PUJO). Glomerular Filtration Rate (GFR) greater than 10 ml/min. Open to both genders.

Exclusion Criteria:

* Active infection. GFR less than 10 ml/min. Presence of a single kidney. Patients with kidney or multiple congenital anomalies. Pregnancy.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2024-10-11 (Actual); Primary Completion 2024-10-11 (Actual); Study Completion 2025-12-04 (Estimated)

PRIMARY OUTCOMES:
Operative Success Rate | 3 days
  evaluating the effectiveness of each surgical method in resolving PUJO

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine Al-Azhar University, Asyut, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Individual Participant Data (IPD) might not be shared due to privacy and confidentiality concerns. The ethical considerations mentioned in the study include informed consent obtained from patients regarding the surgery and data privacy. Sharing IPD could potentially compromise patient anonymity and expose sensitive personal health information, which must be protected under ethical research practices and relevant data protection regulations.

REFERENCES:
- [Background] Bar-Sever Z, Shammas A, Gheisari F, Vali R. Pediatric Nephro-Urology: Overview and Updates in Diuretic Renal Scans and Renal Cortical Scintigraphy. Semin Nucl Med. 2022 Jul;52(4):419-431. doi: 10.1053/j.semnuclmed.2021.12.002. Epub 2022 Jan 11. PMID 35031115